CLINICAL TRIAL: NCT02625272
Title: A Novel Technique of Hand-assisted Laparoscopic Right Hemicolectomy With Complete Mesocolic Excision and Central Vascular Ligation for Right Colon Cancer: A Randomized Controlled Trial
Brief Title: A Novel Technique of HALS With CME and CVL for RCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Chief of Department of Gastrointestinal Surgery, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALS-CME 201512
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Colon Neoplasms
Keywords: hand-assisted laparoscopic surgery; right colon cancer; complete mesocolic excision; no touch isolation; recurrence; overall survival
MeSH Terms: conditions — Colonic Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): The novel hand-assisted laparoscopic surgery with complete mesocolic excision and central vascular ligation for right colon cancer. In this group, greater omentum, transverse colon, and ileum were brought out through the hand-port incision at the beginning of the operation and divided extracorporeally.
  Interventions: Procedure: Group A
- Group B (No Intervention): novel laparoscopic surgery with complete mesocolic excision and central vascular ligation for right colon cancer. In this group, greater omentum, transverse colon, and ileum were divided at the beginning of the operation intracorporeally.
- Group C (No Intervention): the traditional laparoscopic surgery with complete mesocolic excision and central vascular ligation for right colon cancer.

INTERVENTIONS:
Procedure: Group A — The novel hand-assisted laparoscopic surgery with complete mesocolic excision and central vascular ligation for right colon cancer. In this group, greater omentum, transverse colon, and ileum were brought out through the hand-port incision at the beginning of the operation and divided extracorporeally.
  Arms: Group A

SUMMARY:
The purpose of this study is to determine the short and long outcomes of the novel technique of hand-assisted laparoscopic right hemicolectomy with complete mesocolic excision and central vascular ligation for right colon cancer.

DETAILED DESCRIPTION:
Laparoscopic colectomy was first described by Jacobs in the early 1990s. Since then, as a minimally invasive approach, laparoscopic surgery has been gaining popularity for colorectal resection. Compared to open colectomy, laparoscopic colectomy has advantages in blood loss, recovery of bowel function, need for narcotic analgesics, and hospital stay. The long-term outcome of laparoscopic surgery for colon cancer has also been proved.

Complete mesocolic excision (CME) for colon cancer was reemphasized, with the merits of providing better cancer clearance and higher 5 year survival rate. Recently, it has been reported that patients with or without lymph node metastasis both benefit from a wider mesenteric excision including as many negative lymph nodes as possible. The use of D3 lymphadenectomy in colon cancer has been the state of art for decade in Asian countries. A comparison between Japanese D3 resection and European CME with central vascular ligation (CVL) showed that both series were oncologically superior to the traditional right hemicolectomy. Most recently, a consensus is reached between European and Japanese experts that a more radical approach combining CME and D3 lymphadenectomy are oncologically preferable.

Laparoscopic right hemicolectomy with CME or D3 lymphadenectomy have been reported to be feasible and safe by several authors. However, due to the notorious high rate of vascular variations in right colon, laparoscopic right-sided CME with CVL or D3 resection in obese patient remains challenging, even at experienced hands. Two of the major technical difficulties include the identifying of superior mesenteric vein (SMV) in thick layer of fatty tissue and dissection around the middle colic vessels. Here the investigators report a novel technique to tackle these two problems by combining transection of the bowels through the small incision and a medial to lateral approach of hand-assisted laparoscopic (HAL) surgery. The details are as followed:

Surgical Techniques Operation steps outside the abdominal cavity Under general anesthesia, the patient was placed in the supine position with legs split-ted. A middle incision about 7 centimeters long was made around the umbilicus, which was used for placing Lapdisc. This procedure started with transection of great omentum, transverse colon and the distal ileum through the self-expandible Lapdisc.

Transect transverse colon For cancer at ascending colon or cecum, the transverse colon should be divided at a site between the left and right branches of middle colic artery. For hepatic flexural or transverse colon cancer, the transverse colon should be divided at the left side of middle colic artery. After transverse colon was divided, the two ends of transverse colon were returned into the abdomen.

Transect distal ileum Distal ileum was transected 15 to 25 cm from ileocecal valve. After that, the distal end of superior mesenteric vessels were easily identified and severed. By holding the stump, dissection around the superior mesenteric artery (SMA) and SMV could be easily achieved and advanced up to the level of duodenum. And in most cases, the ileocolic artery and vein could be cut at their origins through this small incision. Then, the bowel was returned.

Establish pneumoperitoneum Three trocars were engaged for this procedure: port A was in the left lower quadrant as the main working port; port B was in the upper left quadrant for camera port; and port C was slightly below the xiphoid and used mainly for retracting the mesocolon or the stomach. Next, the Lapdisc was placed and pneumoperitoneum with a pressure of 10-12 mmHg was established.

D3 lymph node dissection with CME and CVL The D3 lymphadenectomy and mobilization of colon were then performed intracorporeally. The course of lymphadenectomy was divided into four steps.

First: Cut peritoneum over SMA and identified the pancreatic neck The surgeon held the middle colic vessels and pulled the mesentery ventrally and finished dividing the mesocolon to ensure a direct view of the pancreatic neck. Open the peritoneum over the SMA and advance cephalad till the pancreas was exposed.

Second: Serving of arterial branches to right colon To identify the arterial branches that cross over the SMV to supply the right sided colon, cares must be taken to take a very thin slice of fat tissue between two blades of Harmonic with the inactive blade facing the SMV, and not to take a big bite of tissue in one time to avoid involving the vessel itself. Before dealing with the middle colic artery, it was better to expose the dorsal edge of pancreatic neck which also marks the anterior level of SMV. Then, both the right colic and middle colic artery were identified. With the help of a finger, it was much easier to push the forcep through behind a vessel and apply ham-locks to the origin of the middle colic artery and the right colic artery. Then the two arteries were divided.

Third: Serving of venous branches from the colon After exposure of the whole length of SMV, the middle colic vein was likely to show itself without much dissection. The middle colic vein was clipped and divided. Then dissect along the right side of SMV. The ileocolic vein had already been divided. The right colic vein, which drains into SMV directly, was clipped and divided. Then dissect along the pancreatic neck.

Fourth: Dissection in front of the pancreatic head. Dissection was continued cephalad, the gastroepiploic vein was observed before dealing with it, and the pancreatic head was exposed. Dissection in front of anterior pancreatoduodenal fascia and blunt dissection was employed for separation mesocolon from the Toldt's fascia.

Mobilization of the right colon With the finger providing constantly changing counter-retraction, the mobilization of mesocolon could be carried out in a fast and precise manner. Mobilizing the cecum from behind the mesocolon called for the surgeon to turn his hand with the palm facing ventrally, and the camera holder turned the camera rod to view mesocolon from behind. Because all the vessels feeding the right sided colon as well as the marginal artery had been severed, the tumor was bloodless during the mobilization of colon. Last, dissect the gastrocolic ligament. For patients with an ascending colon cancer, the gastroepiploic vessels were preserved. With a good retraction provided by hand, the mobilization of mesocolon was an easy task after the medial approach dissection.

Anastomosis After right colon was excised, a side-to-side ileocolic anastomosis was created, and the mesenteric defect was closed extra-corporeally through the small incision.

According to our previous study, this novel HAL right hemicolectomy with CME and CVL is technically feasible and safe. This novel technique carries the merit of blocking all the blood supply to the colon before the mobilization of the tumor and is more in line with the "no touch isolation" technique.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed right colon cancer
* Clinical stage: I, II, III
* No preoperative chemoradiotherapy
* No past surgical history
* No serious preoperative complication
* Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0-1
* Age: 18-80
* Written informed consent

Exclusion Criteria:

* Malignant neoplasm of other sites (including transverse, descending, sigmoid colon cancer, and rectal cancer)
* Metastatic cancer
* Multiple cancer
* Serious complications (including bowel perforation, bowel obstruction, gastrointestinal hemorrhage)
* Pregnant and lactating women
* Psychological disorder
* Steroid administration
* Cardiac infarction within six months
* Severe pulmonary emphysema and pulmonary fibrosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-11 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
operative time | 1 day
the content RNA of CEA and CK20 in circulating tumor cells and ascites | 1 week

SECONDARY OUTCOMES:
postoperative complications | 1 year
overall survival | 3 years
disease-free survival | 3 years
3-year local recurrence | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, MD,PhD, Principal Investigator — West China Hospital
Locations (1):
- West China hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Background] Peters WR, Bartels TL. Minimally invasive colectomy: are the potential benefits realized? Dis Colon Rectum. 1993 Aug;36(8):751-6. doi: 10.1007/BF02048366. PMID 8348865
- [Background] Veldkamp R, Kuhry E, Hop WC, Jeekel J, Kazemier G, Bonjer HJ, Haglind E, Pahlman L, Cuesta MA, Msika S, Morino M, Lacy AM; COlon cancer Laparoscopic or Open Resection Study Group (COLOR). Laparoscopic surgery versus open surgery for colon cancer: short-term outcomes of a randomised trial. Lancet Oncol. 2005 Jul;6(7):477-84. doi: 10.1016/S1470-2045(05)70221-7. PMID 15992696
- [Background] Colon Cancer Laparoscopic or Open Resection Study Group; Buunen M, Veldkamp R, Hop WC, Kuhry E, Jeekel J, Haglind E, Pahlman L, Cuesta MA, Msika S, Morino M, Lacy A, Bonjer HJ. Survival after laparoscopic surgery versus open surgery for colon cancer: long-term outcome of a randomised clinical trial. Lancet Oncol. 2009 Jan;10(1):44-52. doi: 10.1016/S1470-2045(08)70310-3. Epub 2008 Dec 13. PMID 19071061
- [Background] Naitoh T, Gagner M, Garcia-Ruiz A, Heniford BT, Ise H, Matsuno S. Hand-assisted laparoscopic digestive surgery provides safety and tactile sensation for malignancy or obesity. Surg Endosc. 1999 Feb;13(2):157-60. doi: 10.1007/s004649900928. PMID 9918620
- [Background] Meijer DW, Bannenberg JJ, Jakimowicz JJ. Hand-assisted laparoscopic surgery: an overview. Surg Endosc. 2000 Oct;14(10):891-5. doi: 10.1007/s004640020019. PMID 11080398
- [Background] Aalbers AG, Biere SS, van Berge Henegouwen MI, Bemelman WA. Hand-assisted or laparoscopic-assisted approach in colorectal surgery: a systematic review and meta-analysis. Surg Endosc. 2008 Aug;22(8):1769-80. doi: 10.1007/s00464-008-9857-4. Epub 2008 Apr 24. PMID 18437486
- [Background] Chung CC, Ng DC, Tsang WW, Tang WL, Yau KK, Cheung HY, Wong JC, Li MK. Hand-assisted laparoscopic versus open right colectomy: a randomized controlled trial. Ann Surg. 2007 Nov;246(5):728-33. doi: 10.1097/SLA.0b013e318123fbdf. PMID 17968162
- [Background] Kusminsky RE, Boland JP, Tiley EH. Hand-assisted laparoscopic surgery. Dis Colon Rectum. 1996 Jan;39(1):111. doi: 10.1007/BF02048280. No abstract available. PMID 8601348
- [Background] Handoscopic surgery: a prospective multicenter trial of a minimally invasive technique for complex abdominal surgery. Southern Surgeons' Club Study Group. Arch Surg. 1999 May;134(5):477-85; discussion 485-6. PMID 10323419
- [Background] Hohenberger W, Weber K, Matzel K, Papadopoulos T, Merkel S. Standardized surgery for colonic cancer: complete mesocolic excision and central ligation--technical notes and outcome. Colorectal Dis. 2009 May;11(4):354-64; discussion 364-5. doi: 10.1111/j.1463-1318.2008.01735.x. Epub 2009 Nov 5. PMID 19016817
- [Background] Petrovic T, Radovanovic Z, Breberina M, et al. Complete mesocolic excision with central supplying vessel ligation- new technique in colon cancer treatment. Arch Oncol, 2010; 18(3) : 84- 85.
- [Background] West NP, Hohenberger W, Weber K, Perrakis A, Finan PJ, Quirke P. Complete mesocolic excision with central vascular ligation produces an oncologically superior specimen compared with standard surgery for carcinoma of the colon. J Clin Oncol. 2010 Jan 10;28(2):272-8. doi: 10.1200/JCO.2009.24.1448. Epub 2009 Nov 30. PMID 19949013
- [Background] West NP, Morris EJ, Rotimi O, Cairns A, Finan PJ, Quirke P. Pathology grading of colon cancer surgical resection and its association with survival: a retrospective observational study. Lancet Oncol. 2008 Sep;9(9):857-65. doi: 10.1016/S1470-2045(08)70181-5. Epub 2008 Jul 28. PMID 18667357
- [Background] West NP, Kobayashi H, Takahashi K, Perrakis A, Weber K, Hohenberger W, Sugihara K, Quirke P. Understanding optimal colonic cancer surgery: comparison of Japanese D3 resection and European complete mesocolic excision with central vascular ligation. J Clin Oncol. 2012 May 20;30(15):1763-9. doi: 10.1200/JCO.2011.38.3992. Epub 2012 Apr 2. PMID 22473170
- [Background] Feng B, Sun J, Ling TL, Lu AG, Wang ML, Chen XY, Ma JJ, Li JW, Zang L, Han DP, Zheng MH. Laparoscopic complete mesocolic excision (CME) with medial access for right-hemi colon cancer: feasibility and technical strategies. Surg Endosc. 2012 Dec;26(12):3669-75. doi: 10.1007/s00464-012-2435-9. Epub 2012 Jun 26. PMID 22733200
- [Background] Adamina M, Manwaring ML, Park KJ, Delaney CP. Laparoscopic complete mesocolic excision for right colon cancer. Surg Endosc. 2012 Oct;26(10):2976-80. doi: 10.1007/s00464-012-2294-4. Epub 2012 May 2. PMID 22549374
- [Background] Takemasa I, Uemura M, Nishimura J, Mizushima T, Yamamoto H, Ikeda M, Sekimoto M, Doki Y, Mori M. Feasibility of single-site laparoscopic colectomy with complete mesocolic excision for colon cancer: a prospective case-control comparison. Surg Endosc. 2014 Apr;28(4):1110-8. doi: 10.1007/s00464-013-3284-x. Epub 2013 Nov 8. PMID 24202709
- [Background] Storli KE, Sondenaa K, Furnes B, Eide GE. Outcome after introduction of complete mesocolic excision for colon cancer is similar for open and laparoscopic surgical treatments. Dig Surg. 2013;30(4-6):317-27. doi: 10.1159/000354580. Epub 2013 Sep 10. PMID 24022524
- [Background] BARNES JP. Physiologic resection of the right colon. Surg Gynecol Obstet. 1952 Jun;94(6):722-6. No abstract available. PMID 14931182
- [Background] Turnbull RB Jr, Kyle K, Watson FR, Spratt J. Cancer of the colon: the influence of the no-touch isolation technic on survival rates. Ann Surg. 1967 Sep;166(3):420-7. doi: 10.1097/00000658-196709000-00010. No abstract available. PMID 6039601
- [Background] Wiggers T, Jeekel J, Arends JW, Brinkhorst AP, Kluck HM, Luyk CI, Munting JD, Povel JA, Rutten AP, Volovics A, et al. No-touch isolation technique in colon cancer: a controlled prospective trial. Br J Surg. 1988 May;75(5):409-15. doi: 10.1002/bjs.1800750505. PMID 3292002
- [Derived] Yang X, Wu Q, Jin C, He W, Wang M, Yang T, Wei M, Deng X, Meng W, Wang Z. A novel hand-assisted laparoscopic versus conventional laparoscopic right hemicolectomy for right colon cancer: study protocol for a randomized controlled trial. Trials. 2017 Jul 26;18(1):355. doi: 10.1186/s13063-017-2084-3. PMID 28747220